CLINICAL TRIAL: NCT06852430
Title: Factors Associated With Advanced HIV Disease and Poor Nutrition Among People Living With HIV: A Hospital-based Study
Brief Title: Factors Associated With Advanced HIV and Poor Nutrition Among People Living With HIV
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salma Hussein Badry, Doctor, Assiut University
Other Study IDs: Advanced HIV, poor nutrition
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Advanced HIV Disease; Poor Nutriyion Among HIV Patients
Keywords: Advanced HIV disease; AIDS; Acquired immunodeficiency syndrome; Nutrition in HIV disease; People living with HIV; PLWH
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People living with Advanced HIV disease: Factors associated with advanced HIV disease
- People with Early HIV disease: Factors associated with early HIV disease

SUMMARY:
Aim of the work:

1. To determine the frequency of advanced HIV among PLWH in Assiut University Hospital.
2. To assess the nutritional patterns and frequency of poor nutrition among PLWH.
3. To evaluate factors associated with advanced HIV disease and poor nutrition among PLWH.

DETAILED DESCRIPTION:
Human immunodeficiency virus (HIV) is an RNA virus that attacks the human body's immune system, which results, in advanced cases, in expression of opportunistic infections (1). HIV infection represents a global public health burden (2, 3). In Egypt, in 2022, about 34,000 people (<0.1%) were positive for HIV (4). There is 25-30% annual increase of newly confirmed HIV cases in Egypt over the last 10 years (5).

The WHO defines advanced HIV disease as having CD4+ T-cell count <200 cell/mm3 or having an acquired immune deficiency syndrome (AIDS)-related infection (stage 3 or 4 of HIV infection) regardless of the CD4+ T-cell count (1).

The WHO reported, in 2022, that 630,000 people living with HIV (PLWH) died from AIDS-related diseases worldwide (which is 51% fewer than those in 2010) (2, 3, 6). In Egypt, the AIDS-related deaths increased from <100 PLWH in 1990 to <1000 PLWH in 2021 (5).

PLWH are usually malnourished due to opportunistic infections, poor food intake, changes in metabolic activity or chronic illnesses. Malnutrition leads to more impairment of the immune system and further disease progression (7).

According to 2023 Global Hunger index, Egypt is at a moderate level of food insecurity, ranking 57 out of 125 countries. 14.4% of the Egyptian population are food insecure (8).

In Egypt, there is lack of data about the frequency of advanced HIV disease and the nutritional status among PLWH and associated factors. Monitoring these factors could help in early treatment of HIV infection, prevention of further virus transmission and enhancement of the nutritional pattern among PLWH.

ELIGIBILITY:
Inclusion Criteria:

* (1) Newly diagnosed people living with HIV (PLWH), (2) Patients previously diagnosed with HIV but non-compliant to treatment.

Exclusion Criteria:

* (1) PLWH compliant on ART, (2) PLWH who refuse to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People living with HIV disease who attend HIV Counselling Clinic and other departments at Assiut University Hospitals
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-22 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Factors associated with advanced HIV disease and poor nutrition among people living with HIV disease. | Febraury 2025 to December 2026
  To study factors associated with advanced HIV disease and poor nutrition among people living with HIV

CONTACTS AND LOCATIONS:
Overall Officials: Haidi KaramAllah Ramadan, Assisstant professor, Study Director — Assiut University; Ehab Fawzy Abdou, Professor, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Boutros S, Skordis J. HIV/AIDS surveillance in Egypt: current status and future challenges. East Mediterr Health J. 2010 Mar;16(3):251-8. PMID 20795437
- [Result] Rezazadeh L, Ostadrahimi A, Tutunchi H, Naemi Kermanshahi M, Pourmoradian S. Nutrition interventions to address nutritional problems in HIV-positive patients: translating knowledge into practice. J Health Popul Nutr. 2023 Sep 8;42(1):94. doi: 10.1186/s41043-023-00440-z. PMID 37684634
- [Result] Ghazy RM, Al Awaidy S, Taha SHN. Trends of HIV indicators in Egypt from 1990 to 2021: time-series analysis and forecast toward UNAIDS 90-90-90 targets. BMC Public Health. 2023 Apr 1;23(1):625. doi: 10.1186/s12889-023-15490-5. PMID 37005670
- See also: WHO page about HIV, available at: https://www.who.int/news-room/fact-sheets/detail/hiv-aids?gad_source=1&gclid=Cj0KCQjwvb-zBhCmARIsAAfUI2sL_nGP-V-oca55dZe0OroljeQgljfFO5_s1FhbC6xFMxF_mWBCr — https://www.who.int/news-room/fact-sheets/detail/hiv-aids?gad_source=1&gclid=Cj0KCQjwvb-zBhCmARIsAAfUI2sL_nGP-V-oca55dZe0OroljeQgljfFO5_s1FhbC6xFMxF_mWBCrFMaAhNAEALw_wcB
- See also: WHO 2022, available at: https://www.who.int/news-room/fact-sheets/detail/hiv-aids?gad_source=1&gclid=Cj0KCQjwvb-zBhCmARIsAAfUI2sL_nGP-V-oca55dZe0OroljeQgljfFO5_s1FhbC6xFMxF_mWBCr — https://www.who.int/data/gho/data/indicators/indicator-details/GHO/number-of-deaths-due-to-hiv-aids#:~:text=An%20estimated%20380%20000%20%5B300,by%20almost%2056%25%20since%202010